CLINICAL TRIAL: NCT04076150
Title: A First-in-Human Study to Access Feasibility and Safety of the Optimum Aortic Valve Implant
Brief Title: Safety and Performance Study of the Optimum Transcatheter Aortic Valve
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thubrikar Aortic Valve, Inc. (Industry)
Collaborators: KCRI (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: THUB-CLIN-2018-01
Record Dates: First submitted 2019-08-09; First posted 2019-09-03 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Severe Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients Receiving Optimum TAV (Experimental): Patients with symptomatic severe aortic stenosis that will be treated via transcatheter aortic valve implantation procedure
  Interventions: Device: Transcatheter Aortic Valve (TAV) Implantation With The Optimum TAV System

INTERVENTIONS:
Device: Transcatheter Aortic Valve (TAV) Implantation With The Optimum TAV System — Treating patients with severe symptomatic aortic stenosis via transcatheter aortic valve implantation by implanting the Optimum TAV inside the native diseased valve via a the Precision Catheter. The Optimum TAV and Precision Catheter together are the Optimum TAV System.
  Other Names: Transcatheter Aortic Valve Replacement

SUMMARY:
The TAVI (Thubrikar Aortic Valve, Inc.) -1 Study: Safety and Performance Study of the Optimum Transcatheter Aortic Valve- First-in-human study to assess feasibility and safety of the Optimum Aortic Valve Implant

DETAILED DESCRIPTION:
The purpose of the study is to assess the safety and performance of the Optimum TAV (Transcatheter Aortic Valve) in patients with symptomatic, severe aortic stenosis who are deemed high-risk for SAVR (Surgical Aortic Valve Replacement) or have contraindications or deemed inoperable for SAVR.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and capable to provide informed consent;
2. 70 years of age or older;
3. Echocardiographic or hemodynamic based evidence of calcific (senile) aortic stenosis with one of the following: aortic valve Effective Orifice Area (EAO) ≤ 1.0 cm2 or 0.6 cm2/m2, mean aortic valve gradient ≥35 mmHg or peak aortic valve velocity > 4 m/sec.
4. Symptomatology due to native aortic stenosis resulting in a New York Heart Association (NYHA) functional classification of II or greater.
5. Aortic valve annular diameter ≥ 21 and ≤ 23mm measured by MSCT (Multi-Slice Computed Tomography).
6. A STS (Society of Thoracic Surgeons) score ≥ 8; or Logistic EuroScore I ≥ 15; or a determination by the local heart team that the co-morbidities not captured by the STS or EuroScore are expected to increase the operative mortality risk to > 15%.
7. Geographically available and willing to comply with follow up.

Exclusion Criteria:

1. Congenital unicuspid or bicuspid aortic valve;
2. Noncalcified aortic valve;
3. Valve eccentricity (calcific or otherwise) that in the opinion of the investigator could compromise procedural success;
4. Severe (Grade 3 to 4) aortic, mitral, or tricuspid valve regurgitation;
5. Moderate to severe mitral stenosis;
6. Myocardial infarction within the past 30 days*
7. Echocardiographic evidence of intracardiac mass, thrombus or vegetation;
8. LVEF (Left Ventricular Ejection Fraction) < 30%;
9. Severe pulmonary hypertension with pulmonary systolic pressure greater than two-thirds of systemic pressure;
10. Hemodynamic instability requiring inotropic drug therapy within the past 14 days or mechanical support within the past 6 months; *
11. Presence of significant aortic disease such as atheroma, thrombus, or aneurysm which, in the opinion of the investigator, precludes safe implant delivery;
12. Blood dyscrasias defined as: acute leukopenia, acute anemia, acute thrombocytopenia, history of bleeding diathesis or coagulopathy;
13. Patient ineligible for or refuses blood transfusions;
14. Unfavorable peripheral vascular anatomy or disease (e.g. severe obstructive calcification, severe tortuosity or small vessels) that would preclude passage of catheters from the femoral arterial access to the aorta as evidenced by peripheral MSCT;
15. Gastrointestinal bleeding within the past 30 days; *
16. Stroke or transient ischemic attack (TIA) within past 3 months;*
17. Renal insufficiency as demonstrated by a serum creatinine > 3.0 mg/dL;
18. End stage renal disease requiring chronic dialysis;
19. Active infection requiring ongoing treatment;
20. Need for emergent surgery or intervention other than the investigational procedure;
21. Hypersensitivity or contraindication to procedural medication(s) and device material(s) (e.g. titanium, nickel, pork) which cannot be adequately pre-medicated;
22. Life expectancy < 1 year due to non-cardiac co-morbid conditions;
23. Currently participating in any other investigational drug or device study;
24. Patient lacking capacity to provide informed consent (history of any cognitive or mental health status that would interfere with study participation)
25. Subject found to have an International Normalized Ratio (INR) greater than 2.0 right before the procedure.

    * At the time of procedure, if a subject's medical status has changed since enrollment, the subject shall be re-evaluated for eligibility.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-12-18 (Estimated); Study Completion 2027-05-18 (Estimated)

PRIMARY OUTCOMES:
Device Success | 30 days
  Valve deployed from delivery system successfully
Correct Positioning | 30 days
  Deploying a single Optimum TAV in the intended anatomical position and confirming via fluoroscopy as determined by the implanting physician
Intended Performance of Optimum TAV - Leaflet Function | 30 days
  Evaluate leaflet function by assessing the effective orifice area (EOA) (units: cm^2) via echocardiography
Intended Performance of Optimum TAV - mean aortic valve gradient | 30 days
  Evaluate hemodynamics by assessing the mean aortic valve gradient (units: mmHg) via echocardiography
Intended Performance of Optimum TAV - peak aortic valve velocity | 30 days
  Evaluate hemodynamics by assessing the peak aortic valve velocity (units: m/s) via echocardiography
Intended Performance of Optimum TAV - Paravalvular Leak | 30 days
  Evaluate proper valve sealing by assessing paravalvular leak via echocardiography and fluoroscopy. If paravalvular leak is determined, it will be classified as mild, moderate, or severe.

CONTACTS AND LOCATIONS:
Locations (1):
- John Paul II Hospital, Dept. of Interventional Cardiology, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided